CLINICAL TRIAL: NCT04581733
Title: A Phase 3b Single Arm Clinical Study to Evaluate the Efficacy and Safety of MT1621 in Nucleos(t)Ide Treatment Naïve Pediatric and Adolescent Subjects With Thymidine Kinase 2 (TK2) Deficiency
Brief Title: A Study of the Efficacy and Safety of MT1621 in Thymidine Kinase 2 (TK2) Deficiency (Treatment naïve)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Zogenix MDS, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-1621-104
Record Dates: First submitted 2020-09-29; First posted 2020-10-09 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Thymidine Kinase 2 Deficiency
Keywords: TK2; TK2d; mitochondrial disorder; mitochondrial disease; Mitochondria; deoxythymidine/deoxythymidine substrate enhancement therapy; dC/dT; deoxythymidine/deoxythymidine; primary mitochondrial myopathy; mitochondrial depletion syndrome; Muscle weakness; Muscle atrophy; Loss of mobility; Thymidine kinase 2 deficiency
MeSH Terms: conditions — Mitochondrial Diseases; Muscle Weakness; Muscular Atrophy | interventions — Deoxycytidine; Thymidine

STUDY DESIGN:
Intervention Model Description: This is a Phase 3b study. All participants will receive MT1621 up to a target dose of 400 mg/kg/day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Male and female Participants <18 years
  Interventions: Drug: MT1621

INTERVENTIONS:
Drug: MT1621 — All patients will receive MT1621 up to a target dose of 400 mg/kg/day each dC and dT, as tolerated.
  Other Names: Deoxycytidine (dC) and deoxythymidine (dT)

SUMMARY:
This is a Phase 3b, prospective, single-arm, multicenter, open-label treatment study of the efficacy and safety of MT1621 in pediatric and adolescent patients with thymidine kinase 2 deficiency (TK2d). In order to be eligible for this study, participants must have genetic confirmation of TK2d and must not have ever received MT1621 or nucleos(t)ides before entering the study.

DETAILED DESCRIPTION:
Thymidine kinase 2 (TK2) is a protein involved in the normal function of mitochondria. Thymidine kinase 2 deficiency (TK2d) is a form of mitochondrial DNA depletion syndrome and is a very rare inherited genetic disorder. TK2d leads to abnormally low amounts of DNA in mitochondria and because of this defect, the mitochondria are not able to provide the energy that cells need to function properly, which causes severe muscle weakness, along with host of additional symptoms that may involve the respiration, feeding, and ambulation, and can progress until patients lose many of these abilities. There are no FDA-approved medicines to treat TK2d.

MT1621 is a therapy that targets the underlying pathophysiology of TK2d by restoring mitochondrial DNA (mtDNA) replication fidelity. MT1621 consists of a combination of deoxynucleosides (the building blocks of mtDNA) given orally. Deoxynucleoside combination therapy improves nucleotide balance, increases mtDNA copy number, improves cell function, and prolongs life in preclinical models of TK2d.

This is a Phase 3b, prospective, single-arm, multicenter, open-label treatment study to assess the efficacy and safety of MT1621 in treatment naïve pediatric and adolescent subjects <18 years of age with TK2d. The study seeks to enroll approximately 16 subjects globally in this ultra rare disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be aged birth to <18 years of age on the day of consent.
* Diagnosis of TK2 deficiency based on confirmed disease-causing mutation(s) in the TK2 gene.
* Onset of TK2d at ≤12 years of age as defined as the age at which the first TK2d symptom occurred.

Exclusion Criteria:

* Documented clinically significant central nervous system involvement.
* ALT or AST >3 x upper limit of normal and total bilirubin > 2 x ULN or International Normalized Ratio (INR) >1.5.
* EtCO2>45 mmHg if not on ventilatory support
* Current or prior treatment with nucleos(t)ides for TK2d.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects acquiring a Motor Milestone | 12 months
  Proportion of subjects acquiring a motor milestone not present at baseline after 12 months of MT1621 treatment.

SECONDARY OUTCOMES:
Time to Acquisition of a Motor Milestone | 12 months
  Time to Acquisition of a Motor Milestone that was not present at baseline after 12 months of treatment.
Survival | 12 months
  Survival after 12 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273

IPD SHARING:
Plan to Share IPD: No